CLINICAL TRIAL: NCT05094024
Title: Development of Shelf-Stable, Locally-Sourced, Microbiota-Directed Complementary Foods for Children With Undernutrition
Brief Title: Shelf-Stable MDCF-2 for Children With Undernutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR-21019
Record Dates: First submitted 2021-09-21; First posted 2021-10-26 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Central kitchen-prepared MDCF-2 arm (Active Comparator): Children randomized to this arm will receive 25gm of kitchen-prepared version of MDCF-2 twice daily.
  Interventions: Dietary Supplement: Central kitchen-prepared version of MDCF-2
- Ready-to-use supplementary food (RUSF) arm (Experimental): Children randomized to this arm will receive 25g RUSF twice daily.
  Interventions: Dietary Supplement: Ready-to-use supplementary food (RUSF) arm
- Freshly reconstituted MDCF-2 ingredients (Experimental): Children randomized to this arm will receive individually packaged MDCF-2 ingredients, combined into 21.72g servings provided twice daily.
  Interventions: Dietary Supplement: Freshly reconstituted MDCF-2 ingredients
- MDCF-2 shelf-stable foil pouch prototype with green banana powder (Experimental): Children randomized to this arm will receive 21.77gm of shelf-stable foil pouch prototype with green banana powder twice daily.
  Interventions: Dietary Supplement: MDCF-2 shelf-stable foil pouch prototype with green banana powder
- MDCF-2 shelf-stable foil pouch prototype with sweet potato (Experimental): Children randomized to this arm will receive 23.34gm of MDCF prototype with sweet potato twice daily.
  Interventions: Dietary Supplement: MDCF-2 shelf-stable foil pouch prototype with sweet potato

INTERVENTIONS:
Dietary Supplement: Central kitchen-prepared version of MDCF-2 — Kitchen-prepared MDCF-2 containing chickpea flour, peanut flour, soybean flour, green banana pulp, sugar, soybean oil and micronutrient mix. This version of MDCF-2 will be freshly prepared in central kitchens on a daily basis and provided to participants on the same day. Every child in this arm will be offered 25g of the MDCF-2 formulation twice daily.
  Arms: Central kitchen-prepared MDCF-2 arm
Dietary Supplement: MDCF-2 shelf-stable foil pouch prototype with green banana powder — This shelf-stable foil pouch prototype of MDCF-2 contains chickpea flour, peanut flour, soybean flour, green banana powder, sugar, soybean oil and micronutrient mix, prepared by an industry partner following the formulation developed at icddr,b. Every child in this arm will be offered 21.77g of the formulation twice daily.
  Arms: MDCF-2 shelf-stable foil pouch prototype with green banana powder
Dietary Supplement: MDCF-2 shelf-stable foil pouch prototype with sweet potato — This shelf-stable MDCF prototype contains chickpea flour, peanut flour, soybean flour, sweet potato, sugar, soybean oil and micronutrient mix. This version of MDCF-2 will be prepared by an industry partner following the formulation developed at icddr,b. Every child in this arm will be offered 23.34g of the MDCF formulation twice daily.
  Arms: MDCF-2 shelf-stable foil pouch prototype with sweet potato
Dietary Supplement: Freshly reconstituted MDCF-2 ingredients — This version of MDCF-2 is comprised of its individually packaged ingredients. Separate premeasured sachets of chickpea flour, peanut paste, soybean flour, green banana powder, sugar, soybean oil and micronutrient mix will be combined and reconstituted prior to each feeding session. Every child in this arm will be offered 21.72g of the formulation twice daily.
  Arms: Freshly reconstituted MDCF-2 ingredients
Dietary Supplement: Ready-to-use supplementary food (RUSF) arm — Locally-produced ready-to-use supplementary food (RUSF) is used as part of a nutritional program to treat moderate acute malnutrition in children over 6 months-of-age. RUSF is eaten directly from the package with no dilution, mixing or cooking. RUSF contains rice, lentil, powdered low-fat milk, soybean flour, sugar, and micronutrient mix. Every child in this arm will be offered 25g of the formulation twice daily.
  Arms: Ready-to-use supplementary food (RUSF) arm

SUMMARY:
Background: Children with acute malnutrition have immature gut microbial communities compared to age-matched children with healthy growth that can not be repaired by existing therapeutic foods (Subramanian et al., Nature. 2014). Hence, investigators' recent work in Bangladesh has focused on developing Microbiota-Directed Complementary Foods (MDCF) containing locally-available food ingredients, that repair the gut microbiota of children with acute malnutrition to a configuration that resembles that of healthy children living in the same urban community (Raman et al., Science 2019; Gherig et al., Science 2019).

The investigators recently completed a randomized, controlled proof-of-concept (POC) study of current lead microbiota-directed complementary food, MDCF-2 compared to a standard ready-to-use supplementary food (RUSF), in Bangladeshi children with moderate acute malnutrition (MAM)(Chen et al., N Engl J Med 2021). Children who received MDCF-2 for 3 months exhibited significantly greater repair of their gut microbial communities and faster rates of ponderal growth compared to those treated with RUSF (a formulation that was not designed based on knowledge of its effects on the gut microbiota). The superior effect of MDCF-2 on gut microbiota repair and weight gain was even more notable as the RUSF was significantly more energy dense than MDCF-2.

In the aforementioned POC study, MDCF-2 was prepared fresh daily in icddr,b field kitchens prior to distribution and supervised administration to study participants. The lack of a shelf-stable, bio-equivalent formulation of MDCF-2 limits the ability to perform larger studies in Bangladesh as well as in other geographic settings. This pre-POC study in Bangladeshi children with MAM will assess the bioequivalence of MDCF prototypes that the investigators have developed with the potential for improved storage stability compared to current MDCF-2, using the degree of microbiota repair after 4-weeks of treatment as the primary outcome.

Objective: To develop a scalable, shelf-stable formulation that is bioequivalent to MDCF-2 with respect to microbiota repair in 8-12 month-old Bangladeshi children with MAM after 4-weeks of treatment.

Methods: A 5-arm, randomized single-blind pre-POC study will be conducted in 8-12-month-old Bangladeshi children with MAM to compare the efficacy of alternative MDCF formulations in repairing their gut microbiomes compared to the repair produced by the current kitchen prepared MDCF-2 formulation.

Arm 1 - Reference control: kitchen-prepared MDCF-2

Arm 2 - Ready-to-use supplementary food

Arm 3 - Individually packaged, pre-measured sachets of MDCF-2 ingredients, combined and reconstituted in the home setting prior to consumption.

Arm 4 - MDCF-2 shelf-stable foil pouch formulation with green banana powder.

Arm 5 - MDCF shelf-stable foil pouch formulation with sweet potato instead of green banana.

DETAILED DESCRIPTION:
Study site: The study will be conducted among residents of an under slum community in Baoniabad of Mirpur, one of the 21 administrative units of the nation's capital, Dhaka. Mirpur is selected as the study site because it is inhabited by poor and lower middle-class families, residential and sanitary conditions are typical of any congested urban settlement. Additionally, the investigators have established several field sites in the area and they have ongoing research activities in the community.

Enrollment: A trained Field Research Assistant (FRA) will explain the study in detail, answer any questions from the parent(s), and invite the parent(s) to enrol the child in the study. If the parent(s) are interested to volunteer in the study, the designated staff will proceed to screening and consenting. Screening will consist of a review of the inclusion and exclusion criteria listed above. If the subject is eligible to participate, the process will proceed to consenting consisting of a thorough review of the written consent form in a manner appropriate for the child's parents' literacy level. Prior to signing the consent form, the parents of the participants will have an opportunity to ask any questions about the study. If the FRA determines that participants have demonstrated adequate comprehension of the study, the consent form will be signed by the FRA and the child's parent(s). If the parent(s) are not sufficiently literate to read and/or sign the consent form, consenting and a thumbprint signature will be obtained in the presence of a witness who is not associated with the study. The child's parent(s) will be provided with a copy of the signed consent form.

Children will undergo thorough clinical assessment and laboratory tests (if needed) to exclude any organic diseases or any other causes of secondary malnutrition. Detailed inclusion/exclusion criteria are provided separately below.

At the beginning of the study, information will be collected on the demographic characteristics of the participants (family income, standard/type of housing, family structure, parental education, etc.). FRAs will collect anthropometry data by recording the child's weight using a digital scale with 2 g precision (Seca, model 728, Germany), length (using infantometer, Seca, model 416, Germany), and mid-upper arm circumference (MUAC) to the nearest millimeter (using a non-stretch tape). Collection of anthropometric data will subsequently occur at weekly intervals throughout the study.

Study Design: The study will be 8 weeks in duration and comprise 5 arms, with a minimum of 23 children per arm required to complete the study. Children will be randomly assigned to one of the five arms using a computer generated randomization scheme. Efforts will be made to balance arms with respect to gender. Mothers/primary caregivers will be be advised to maintain their child's current dietary and breastfeeding practices throughout the study. Following a 2-week 'run-in' phase with weekly fecal sample collection and a blood draw, treatment will be initiated. The treatment phase will be for 4 weeks, during which time each test product will be administered at the test center twice daily, separated by at least 6 hours. The amount of each serving actually ingested will be calculated by subtracting the leftover amount from the offered amount. Pre-weighed napkins will be provided; any food that is regurgitated, vomited or spilled will be swabbed, weighed and subtracted from the amount offered. Fecal samples will be collected weekly using established SOPs for rapid cryopreservation. A second blood draw will be performed at the end of the 4-week intervention period. There will be a 2- week post intervention phase during which 2 additional fecal samples will be collected (at the end of weeks 7 and 8) to assess changes in the microbiota that occur after cessation of treatment.

Children will be monitored daily by trained FRAs for any side effects/adverse events (e.g. rash, urticaria due to food allergy, or any significant changes in clinical status). If any adverse events are observed, children will be treated using appropriate management practices at Dhaka Hospital.

Fecal sample collection: Fecal samples will be collected weekly from each study participant during the course of the 8-week study, including during the 2 weeks prior to treatment, the four weeks of treatment, and the two weeks following cessation of treatment (11 samples/ child). Fecal samples will be used for culture-independent analysis of microbial composition using existing SOPs, and for subsequent culture-based initiatives to characterize growth promoting bacterial taxa (Raman et al., Science 2019, 365, eaau 4735; Gehrig et al., Science 2019; 365, eaau4732).

Blood sample collection: 5 mL of blood will be collected from each child immediately prior to initiating treatment, and just after the 4-week period of treatment is complete. Plasma will be prepared immediately and frozen at -80C prior to proteomics analysis as previously described (Gehrig et al., Science 2019, 365, eaau4732; Chen et al., N Engl J Med 2021; 384:1517-1528). Additionally, status of different blood biomarkers (hormonal regulators of appetite and satiety, micronutrient status, and systemic inflammation) will also be assessed using the samples collected before and after the intervention

Sample size estimate: The estimate is informed by fecal 16S rDNA datasets generated in a recent POC study in 12 to 18-month-old Bangladeshi children with moderate acute malnutrition (MAM) who had been treated with the ("reference") kitchen-prepared MDCF-2 formulation. This formulation repaired the microbiota of these children and produced an improvement in the rate of ponderal growth that was superior to that produced by the control Ready-to-Use Supplementary Food (RUSF; Chen et al., 2021). In this POC study, the investigators identified 209 bacterial taxa (Amplicon Sequence Variants; ASVs) that were present above 5 counts in at least 5% of the 939 fecal samples analyzed from 118 participants (Chen et al., 2021).

The investigators calculated 95% confidence intervals (CI; mean ± 1.96 standard error) for the change (delta) in abundance of each of the 209 bacterial taxa ASVs between day 0 (pre-intervention) and 4 weeks of intervention for the 59 children who completed treatment in the MDCF-2 group of the POC study. The investigators used a bootstrapping approach with ASV data from 5000 subsets of children from the MDCF-2 group and 5000 subsets of children from the RUSF group and identified 121 ASVs whose mean changes in abundance fell within the 95% CI of the mean changes for the MDCF-2 participants, but not in children that had received RUSF, with 80% power using a subset (sample) size of 20 children per group ("MDCF-2-responsive ASVs"). Therefore, we will aim to have a minimum of 20 children per arm complete this pre-POC study. Taking into account potential drop-outs (15%), a minimum of 23 children will be recruited per arm.

Analysis plan: To assess the comparability of microbiota repair elicited by alternative/shelf-stable test formulations of MDCF-2 and the reference kitchen-prepared formulation described in Chen et al (2021), the investigators sequence PCR amplicons generated from bacterial 16S rDNA genes present in DNA isolated from fecal samples collected from participants in the different study arms immediately prior to intervention (day 0) and at the end of intervention (day 28). ASV data will be processed using DADA2 (Callahan et al., 2016) and filtered as described in Chen et al. (2021). Using the same approach used for the POC study above, the investigators will calculate 95% confidence intervals of the mean change in abundance of each of the MDCF-2-responsive ASVs identified in this study, between day 0 and day 28, in children who received the reference MDCF-2 formulation, as well as the mean change for each of these ASVs in participants receiving the test formulations.

A test formulation will be considered comparable in efficacy to the reference kitchen-prepared MDCF-2 if >70% of the MDCF-2-responsive ASVs identified in this study have mean changes in abundance (day 0 to day 28) for the test formulation that fall within the 95% CI of their mean changes in abundance in the reference MDCF-2 arm over the same time period. Another embodiment of the analysis of microbial community repair elicited by the reference MDCF-2 and test formulations will involve a comparison of their respective effects after 4 weeks of treatment on the abundances of metagenome-assembled genomes (MAGs) identified by shotgun sequencing of the same fecal DNA samples used to produce 16S rDNA amplicons.

Exploratory outcomes will include the effects of the test formulations on features of the plasma and fecal proteomes, including MDCF-2-responsive proteins that are associated with various facets of healthy growth, CNS development and immune function, using approaches described in Chen et al., 2021.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) willing to sign consent form
* Child aged 8-12 months
* WLZ score <-2 to -3 without bilateral pedal edema at the time of randomization
* Parent(s) willing to bring the child to the feeding centre according to the pre-defined schedule

Exclusion Criteria: Meeting any of the following criteria will exclude a subject from study participation -

1. Medical conditions: Malnourished children with complications requiring acute phase treatment in a hospital, children with tuberculosis (diagnosis based on WHO 2014 guidelines which have been incorporated in the national TB control guidelines of Bangladesh). The guidelines depend upon the following five diagnostic principles (three out of five should be positive):

   * Specific symptoms of TB
   * Specific signs of TB
   * Chest X-ray
   * Mantoux test
   * History of contact
2. Any congenital/acquired disorder affecting growth, i.e., known case of trisomy-21 or cerebral palsy; children on an exclusion diet for the treatment of persistent diarrhea; having known history of soy, peanut or milk protein allergy
3. Severe anemia (< 8 mg/dl)
4. Antibiotic use (within last 15 days before the onset of intervention)
5. Ongoing maternal antibiotic usage for breastfeeding infants
6. Receiving concurrent treatment for another condition

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2021-10-31 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Equivalence in the response to MDCF-2 and a test MDCF formulation, based on the change in representation of gut bacterial taxa after 4-weeks of treatment with MDCF-2, compared to the change after treatment with the test MDCF for 4-weeks. | Baseline to 4-weeks of treatment.
  V4-16S rDNA amplicons and shotgun sequencing datasets will be generated from fecal samples collected from each child in each group prior to, during, and after treatment to determine the abundances of MDCF-2 responsive bacterial taxa.
  Equivalence will be defined as the absence of a statistically significant difference after 4-weeks of treatment in the representation of fecal bacterial taxa associated with the response to MDCF-2 in participants receiving a test MDCF, compared to the representation of these bacterial taxa in participants after receiving the reference MDCF-2 formulation for 4-weeks.

OTHER OUTCOMES:
Changes in the abundances of 7000 circulating plasma proteins | Baseline to end of Week 4
  To expand our understanding of the biological pathways underlying growth impairment in children with MAM and its repair by MDCF-2, plasma proteins will be analyzed using SomaScan- based measurements.
Changes in the concentrations of fecal protein biomarkers of gut inflammation | Baseline to end of Week 4
  To expand our understanding of the biological pathways underlying growth impairment in children with MAM and its repair by MDCF-2, fecal proteins will be analyzed using ELISA based measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Mirpur, Dhaka, Bangladesh

REFERENCES:
- [Result] Raman AS, Gehrig JL, Venkatesh S, Chang HW, Hibberd MC, Subramanian S, Kang G, Bessong PO, Lima AAM, Kosek MN, Petri WA Jr, Rodionov DA, Arzamasov AA, Leyn SA, Osterman AL, Huq S, Mostafa I, Islam M, Mahfuz M, Haque R, Ahmed T, Barratt MJ, Gordon JI. A sparse covarying unit that describes healthy and impaired human gut microbiota development. Science. 2019 Jul 12;365(6449):eaau4735. doi: 10.1126/science.aau4735. PMID 31296739
- [Result] Gehrig JL, Venkatesh S, Chang HW, Hibberd MC, Kung VL, Cheng J, Chen RY, Subramanian S, Cowardin CA, Meier MF, O'Donnell D, Talcott M, Spears LD, Semenkovich CF, Henrissat B, Giannone RJ, Hettich RL, Ilkayeva O, Muehlbauer M, Newgard CB, Sawyer C, Head RD, Rodionov DA, Arzamasov AA, Leyn SA, Osterman AL, Hossain MI, Islam M, Choudhury N, Sarker SA, Huq S, Mahmud I, Mostafa I, Mahfuz M, Barratt MJ, Ahmed T, Gordon JI. Effects of microbiota-directed foods in gnotobiotic animals and undernourished children. Science. 2019 Jul 12;365(6449):eaau4732. doi: 10.1126/science.aau4732. PMID 31296738
- [Result] Subramanian S, Huq S, Yatsunenko T, Haque R, Mahfuz M, Alam MA, Benezra A, DeStefano J, Meier MF, Muegge BD, Barratt MJ, VanArendonk LG, Zhang Q, Province MA, Petri WA Jr, Ahmed T, Gordon JI. Persistent gut microbiota immaturity in malnourished Bangladeshi children. Nature. 2014 Jun 19;510(7505):417-21. doi: 10.1038/nature13421. Epub 2014 Jun 4. PMID 24896187
- [Result] Chen RY, Mostafa I, Hibberd MC, Das S, Mahfuz M, Naila NN, Islam MM, Huq S, Alam MA, Zaman MU, Raman AS, Webber D, Zhou C, Sundaresan V, Ahsan K, Meier MF, Barratt MJ, Ahmed T, Gordon JI. A Microbiota-Directed Food Intervention for Undernourished Children. N Engl J Med. 2021 Apr 22;384(16):1517-1528. doi: 10.1056/NEJMoa2023294. Epub 2021 Apr 7. PMID 33826814
- [Result] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Derived] Mostafa I, Fahim SM, Das S, Gazi MA, Hasan MM, Saqeeb KN, Mahfuz M, Lynn HB, Barratt MJ, Gordon JI, Ahmed T. Developing shelf-stable Microbiota Directed Complementary Food (MDCF) prototypes for malnourished children: study protocol for a randomized, single-blinded, clinical study. BMC Pediatr. 2022 Jul 1;22(1):385. doi: 10.1186/s12887-022-03436-6. PMID 35778675